CLINICAL TRIAL: NCT00995254
Title: Reducing Secondhand Smoke Exposure Among Young Children
Brief Title: Secondhand Smoke Exposure Reduction Among Young Children in China
Acronym: China SHARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Abu S Abdullah, Boston University School of Public Health
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 072223_CIA
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Secondhand Smoke Exposure; Respiratory Illness; Smoking Cessation
Keywords: secondhand smoke; children; Chinese; respiratory symptoms; household smoking policy; Respiratory illnesses among children
MeSH Terms: conditions — Smoking Cessation; Signs and Symptoms, Respiratory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control group will ONLY receive SHI after completion of the study
- Intervention group (Experimental): Intervention group will receive smoking hygiene intervention (SHI) at three individualized contacts.
  Interventions: Behavioral: SHI counseling

INTERVENTIONS:
Behavioral: SHI counseling — The SHI will be delivered in three different individualized counseling sessions: the initial in person counseling (30-45 minutes), at 1 week in person or telephone counseling (15-30 minutes) and at 1 month in person counseling (15-30 minutes). During the initial counseling, CHWs will emphasize the health hazards of SHS exposure towards young children and its possible illness outcomes. Then subjects will be asked to assess the SHS exposure of children in the household (e.g., estimating the number of hours for SHS exposure on the child per week or day) and the source of SHS. The concept of smoking hygiene and non-smoking household policy will be discussed and any potential barriers ascertained. Furthermore, the CHWs will use the transtheoretical model of Prochaska to assess the stage of readiness of the household member to change smoking behavior existing in the household. Individuals who wish to quit smoking will receive a brief advice on quitting smoking.
  Arms: Intervention group

SUMMARY:
Second hand smoking (SHS) is a health hazard to infants and children, in whom it is associated with lower respiratory tract infections, wheezing, cough, middle ear infections and sudden infant death syndrome. Evidence from developed nations suggests that measures to reduce exposure to SHS can improve children's health outcomes; this has not been systematically studied in a developing country setting. The investigators hypothesize that implementation of a package of smoking hygiene intervention measures delivered by community health workers (CHWs) will reduce Chinese children's exposure to SHS and improve their respiratory health.

To test this hypothesis, the investigators have identified three specific aims: (1) to obtain baseline data on second hand tobacco exposure among young children, health status of young children and smoking status of parents and other household members, (2) to generate preliminary effectiveness data for CHW-delivered SHI, and (3) to develop culturally appropriate biochemical measures to assess children's exposure to household SHS. The investigators propose to conduct this study in an urban district in Shanghai, China. After an initial assessment, the investigators will conduct a randomized controlled trial of households in a community, selected based on important study criteria, within the district. The investigators selected this design because it is most likely to produce a scientifically valid answer to our primary study question. All eligible smokers in the intervention group will receive behavioral counseling to address health hazards of SHS towards children, brief advice to quit or to adopt a no smoking policy around children, and educational pamphlets on the hazards of SHS, from a trained CHW in their community. A questionnaire will be used for data collection at the start and at 2 and 6 months. To assess the extent of total SHS exposure, children's urine cotinine (the indicator of nicotine) level will be measured at the first contact and at 2-and 6- months. To validate household members reported level of smoking the investigators will measure air nicotine levels of a sub-sample (10%) of households via passive monitors. The results of this study will provide clinical evidence for the development of CHW-delivered interventions designed to reduce exposure to SHS and improve the respiratory health of children in a resource-poor community. If successful, the program can serve as a model for implementation in other developing country settings. Furthermore, successful results could also be used to draft guidelines for health promotion interventions, which could be implemented as a policy for all primary health care settings. Finally, the study, which would be the first of its type in a developing country setting, will form the basis for future research and program development in the area of SHS.

ELIGIBILITY:
Inclusion Criteria:

1. household member has smoked one or more cigarettes daily for the past 30 days as self reported;
2. household smoker smokes a total of at least 10 cigarettes per week at home in the presence of the child, as self reported;
3. smoker household member and the child are living together in the same household and will live together during the entire period of the study;
4. residents of the study community;
5. able to communicate in Mandarin Chinese or local Shanghai dialect; AND
6. has signed an informed consent form or given verbal consent (for those who cannot read and write).

Exclusion Criteria:

1. reported residential coal burning and confirmed by the interviewer;
2. households with breast-feeding child;
3. household members do not smoke at home;
4. smoker member does not live in the same household as the under 5 child;
5. non-local community resident; OR
6. not able to communicate in Mandarin Chinese or Shanghai dialect.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
improvement of smoking hygiene practices within the household as reported by the subjects (i.e. reduction in the number of cigarettes smoked indoors at home while a child was present during the previous week) | at 6 month follow up

SECONDARY OUTCOMES:
reduction of respiratory illness incidence among young children as reported by key household members | at 6 month follow up
reduction of reported health care utilization due to respiratory disease | at 6 months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health Centers, Shanghai, Shanghai Municipality, China